CLINICAL TRIAL: NCT01561833
Title: A Pilot Study of Sorafenib Examining Biomarkers in Refractory or Relapsed T-Cell Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901004690
Record Dates: First submitted 2012-03-13; First posted 2012-03-23 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-03

CONDITIONS: T Cell Lymphoma
Keywords: relapsed or refractory T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Recurrence | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Sorafenib, 400 mg PO twice daily
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Intrapatient dose reduction to 400 mg once daily and then 400 mg every other day will be allowed depending on the type and severity of toxicity encountered provided that criteria for patient withdrawal from study treatment have not been met.

SUMMARY:
This study will be a pilot study of sorafenib 400mg PO twice daily in refractory T-cell lymphomas including peripheral T-cell lymphoma (PTCL), angioimmunoblastic lymphadenopathy (AILD), cutaneous T cell lymphoma (CTCL), anaplastic large cell lymphoma (ALCL) and other transformed T-cell lymphomas with the primary objective of studying the biological effects of the multikinase inhibitor, sorafenib.

DETAILED DESCRIPTION:
Primary objectives:

• To study the biological effects of sorafenib 400mg BID on the mitogen-activated protein kinase (MAPK) pathway, specifically the inhibition of extracellular signal-regulated kinases (ERK) phosphorylation, and to correlate with clinical activity in patients with T-cell lymphoma.

Secondary objectives:

* To observe the clinical activity of sorafenib 400mg BID by determining response rate, and progression free survival in patients with T-cell lymphoma. Duration of response and duration of stable disease will also be measured.
* To determine the tolerability of sorafenib in patients with T-cell lymphoma.

Exploratory objectives:

* To observe the effects of sorafenib on T-cell subsets (CD4/CD8 ratio, and Tregs), and the effects of sorafenib on the monocytoid population.
* To observe the effects of sorafenib on the serum cytokine profile.
* To observe the effects of sorafenib on the T-cell receptor pathway, i.e. Lck, ZAP-70, and Syk.
* To observe changes in lymph node or skin morphology including tumor cell infiltrate, vasculature, and the tumor microenvironment in patients treated with sorafenib by performing serial biopsies of lymph nodes or skin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed T-cell lymphoma including PTCL, AITL, CTCL, ALCL (Alk+, and Alk-), and other transformed T-cell lymphomas
* Age > 18 years old
* Measureable disease, as defined by the Cheson criteria
* ECOG Performance Status of 0 or 1
* Life expectancy > 12 weeks
* Adequate bone marrow, liver and renal function
* Patients with hemoglobin < 8.5g/dL, or ANC 500-1000/mm3, or platelets 50,000-75,000/mm3 (Grade 3), whose cytopenias are due to bone marrow involvement by T-cell lymphoma will also be eligible

Exclusion Criteria:

* Prior treatment with sorafenib, or other agents with similar activity, i.e. bevacizumab, imatinib, sunitinib.
* Prior treatment with allogeneic stem cell transplant
* Cardiac disease: Congestive heart failure > class II NYHA.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorafenib
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 12
Age, Customized [Mean (Inter-Quartile Range); unit: years] — Age in years
  years
    Age | 68 [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate to sorafenib. Complete response by recist criteria was complete disappearance of all tumor lesions. partial response was 30% reduction in all sites of disease.
Time Frame: 29 days
Population: all patients enrolled were assessed for response
Measure: Number; unit: participants
Groups:
- Sorafenib: sorafenib
Arm/Group | Sorafenib
Number analyzed (Participants) | 12
participants | 5

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No